CLINICAL TRIAL: NCT02712398
Title: A Prospective, Multi-center Trial of a Long-term Bio-Absorbable Mesh With Sepra Technology in Challenging Laparoscopic Ventral or Incisional Hernia Repair
Brief Title: A Prospective Trial of a Bio-absorbable Mesh in Challenging Laparoscopic Ventral or Incisional Hernia Repair
Acronym: ATLAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DVL-HE-017
Record Dates: First submitted 2016-03-15; First posted 2016-03-18 (Estimated); Results first posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2020-12

CONDITIONS: Hernia, Ventral; Incisional Hernia
MeSH Terms: conditions — Hernia, Ventral; Incisional Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Phasix™ ST (Experimental): Subjects treated with Phasix™ ST mesh
  Interventions: Device: Phasix™ ST

INTERVENTIONS:
Device: Phasix™ ST — Phasix™ ST is a fully resorbable mesh with a hydrogel coating that is also resorbable.

SUMMARY:
The objective of this study is to collect additional data on safety, performance and effectiveness of Phasix™ ST in subjects receiving laparoscopic ventral or incisional hernia repair at high risk for surgical site occurrence (SSO).

DETAILED DESCRIPTION:
Subjects at high risk are defined as having 1 or more of the following co-morbid conditions: body mass index (BMI) between 30-40 kg/m2, inclusive, active smokers, chronic obstructive pulmonary disease (COPD), diabetes, immunosuppression, coronary artery disease, chronic corticosteroid use, low pre-operative serum albumin, advanced age, or renal insufficiency.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 years of age or older
* Subject must be willing to give written informed consent
* Subject must be diagnosed with ventral or abdominal incisional hernia
* Subject must be willing to undergo laparoscopic hernia repair using intraabdominal placement (with or without Component Separation Technique (CST))
* Surgeon must be able to fully close the hernia defect. Defect closure is defined as complete reapproximation of fascial edges, leaving no gap. Since the safety and effectiveness of Phasix™ ST Mesh in bridging repairs has not been evaluated or established, the defect should be closed prior to mesh use.
* Subject is expected to meet the criteria for a Class I wound
* Subjects must have 1 or more of the following pre-study conditions:

  1. Body Mass Index (BMI) between 30-40 kg/m2, inclusive
  2. Active smoker (including if attempts to quit smoking within two weeks of surgery have failed and the patient is still an active smoker at the time of surgery)
  3. COPD presence on patient self-report
  4. Diabetes mellitus (if yes, diagnosis to be confirmed via medical records or laboratory results according to 2014 Joslin Clinical Guideline for Adults with Diabetes)(Appendix 5)
  5. Immunosuppression
  6. Coronary Artery Disease
  7. Chronic corticosteroid use: greater than 6 months systemic use
  8. Serum albumin less than 3.4 g/dL
  9. Advanced age: 75 years or older
  10. Renal insufficiency, defined as serum creatinine concentration ≥2.5 mg/dL

Exclusion Criteria:

* Subject has had 4 or more previous hernia repairs (of the index hernia)
* Subject's hernia is > 350 cm2
* Complete removal of existing mesh from a prior hernia repair (in the same affected area) is not possible
* Subject has intact permanent mesh adjacent to the current hernia to be repaired
* Preperitoneal placement of mesh
* The subject is known to have a collagen disorder
* The subject has peritonitis
* The subject is on or suspected to be placed on chemotherapy medications during any part of the study
* The subject's Body Mass Index (BMI) is > 40 kg/m2
* The subject has cirrhosis of the liver and/or ascites
* Subject is American Society of Anesthesiology Class 4 or 5
* Subject has a life expectancy of less than 2 years at the time of enrollment
* Subject has any condition that, in the opinion of the Investigator, would preclude the use of the study device, or preclude the subject from completing the follow-up requirements
* Subject has a surgical wound classified as Class II (Clean-Contaminated), Class III (Contaminated) or Class IV (Dirty-Contaminated)
* Subject has an active or latent systemic infection
* Patient has a contraindication to placement of mesh
* Subject requires surgical bridge repair as the sole repair
* Subject is pregnant or has plans to become pregnant during the study period
* Subject has enrolled in another interventional clinical study within the last 30 days
* Subject is part of the site personnel directly involved with this study
* Subject has a known allergy to the test device or component materials (patients with known allergies to tetracycline hydrochloride or kanamycin sulfate should be avoided).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Hope, MD, Principal Investigator — New Hanover Regional Medical Center
Locations (16):
- United States (16):
  - Yale-New Haven Medical Center, New Haven, Connecticut
  - Florida Hospital, Celebration, Florida
  - Emory University, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Via-Christi Hospital, Wichita, Kansas
  - Georgetown Community Hospital, Georgetown, Kentucky
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Our Lady of the Lake Regional Medical Center, Baton Rouge, Louisiana
  - Washington University, St Louis, Missouri
  - Methodist Hospital, Omaha, Nebraska
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - Legacy Emanuel Hospital, Portland, Oregon
  - Hershey Penn State Medical Center, Hershey, Pennsylvania
  - Carilion Clinic, Roanoke, Virginia
  - Overlake Hospital, Bellevue, Washington
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phasix™ ST
Started | 120
Completed | 83
Not Completed | 37
Not completed — Withdrawal by Subject | 6
Not completed — Lost to Follow-up | 6
Not completed — Sponsor Decision | 1
Not completed — Physician Decision | 1
Not completed — Death | 2
Not completed — Re-operation | 21

BASELINE CHARACTERISTICS:
Arm/Group | Phasix™ ST
Number analyzed (Participants) | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 84
  >=65 years | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.0 (14.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 119
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 110
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 120
BMI [Mean (Standard Deviation); unit: kg/m^2] | 33.2 (4.48)

OUTCOME MEASURES:

1. Primary Outcome: Surgical Site Occurrence Rate
Description: Proportion of subjects with Surgical Site Occurrences(SSO), which are defined as hematoma, seroma, surgical site infection, wound dehiscence, skin necrosis and fistula requiring intervention. Occurrences at the surgical site will be assessed by physical examination at each study visit through 45 days.
Time Frame: 45 Days
Measure: Number; unit: subjects
Arm/Group | Phasix™ ST
Number analyzed (Participants) | 120
subjects | 1

2. Secondary Outcome: Surgical Site Occurrence Rate
Description: Number of subjects with Surgical Site Occurrences, which are defined as hematoma, seroma, surgical site infection, wound dehiscence, skin necrosis and fistula requiring intervention. Occurrences at the surgical site will be assessed by physical examination at each study visit through 3 months.
Time Frame: 3 months
Measure: Number; unit: subjects
Arm/Group | Phasix™ ST
Number analyzed (Participants) | 120
subjects | 0

3. Secondary Outcome: Hernia Recurrence Rate
Description: Proportion of subjects with hernia recurrence. Hernia recurrence rates will be assessed by physical examination (or if standard of care via CT/MRI or ultrasonography) at each study visit through 24 months. A recurrent hernia will be defined as any hernia identified or confirmed by the investigator, during any study follow-up visit, in approximately the same position as the hernia repaired in the study procedure.
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Phasix™ ST
Number analyzed (Participants) | 120
Participants | 38

4. Secondary Outcome: Pain Visual Analog Scale
Description: Mean change in self-reported pain measured on a Visual Analog Scale between Baseline and 24-month through follow up. Scores are measured on a 10.0 cm line, scores range from 0 to 10, higher values correspond with higher pain perception. The outcome measure is presented as the absolute difference between the pain perception at Baseline and the pain perception at 24-month follow up.
Time Frame: 24 Months
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Phasix™ ST
Number analyzed (Participants) | 120
centimeters | 0.94 (1.63)

5. Secondary Outcome: Device-related Adverse Event Incidence
Description: Proportion of subjects with Investigator-determined device-related adverse events
Time Frame: 24 Months
Measure: Number; unit: subjects
Arm/Group | Phasix™ ST
Number analyzed (Participants) | 120
subjects | 49

6. Secondary Outcome: Rate of Reoperation Due to Index Hernia Repair
Description: Rate of reoperation due to the index hernia repair
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Phasix™ ST
Number analyzed (Participants) | 120
Participants | 22

7. Secondary Outcome: Change in Carolinas Comfort Scale
Description: Each scale score (sensation of mesh, pain or movement limitations) ranges from 0-5 and is the average across the domains. The Total CCS Score ranges from 0-5 and is the average of the 3 scale scores. Low scores represent fewer symptoms or difficulties.
  Absolute values of the Total CCS Score at Baseline, 1-Month follow-up, at 3-Month follow-up, at 6-Month follow-up, at 12-Month follow-up, at 18-Month follow-up, and at 24-Month follow up are reported.
  The absolute value at Baseline, or a change in self-reported quality of life measured by Carolinas Comfort Scale® cannot be reported, as subjects had incorrectly answered the questions on Sensation of Mesh at Baseline where no Phasix Mesh was yet implanted, thereby creating a bias in the results.
Time Frame: 24 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phasix™ ST
Number analyzed (Participants) | 120
units on a scale
  Total CCS Score - Baseline | 1.15 (1.059)
  Total CCS Score - 1 Month | 0.85 (0.938)
  Total CCS Score - 3 Month | 0.34 (0.601)
  Total CCS Score - 6 Month | 0.22 (0.523)
  Total CCS Score - 12 Month | 0.13 (0.353)
  Total CCS Score - 18 Month | 0.17 (0.377)
  Total CCS Score - 24 Month | 0.17 (0.425)

8. Secondary Outcome: Change in SF(Short-form)-12
Description: The Short Form (SF)-12 version 2 (v2) is a multi-purpose, twelve item health survey that measures seven domains of health: general health, physical functioning, role limitations due to physical health (role-physical), role limitations due to emotional problems (role-emotional), bodily pain, vitality and mental health and social functioning. The SF-12v2 yields scale scores for each of these seven health domains, and two summary measures of physical and mental health: the physical component summary (PCS) and mental component summary (MCS). The scores range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
  Absolute values of the PCS and MCS scores at Baseline, 1-Month follow-up, at 3-Month follow-up, at 6-Month follow-up, at 12-Month follow-up, at 18-Month follow-up, and at 24-Month follow up are reported.
Time Frame: 24 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phasix™ ST
Number analyzed (Participants) | 120
score on a scale
  PCS - Baseline | 44.38 (9.635)
  PCS - 1 Month | 40.35 (9.349)
  PCS - 3 Month | 48.83 (8.026)
  PCS - 6 Month | 49.99 (8.277)
  PCS - 12 Month | 50.10 (8.248)
  PCS - 18 Month | 50.48 (8.794)
  PCS - 24 Month | 48.02 (9.739)
  MCS - Baseline | 53.47 (9.493)
  MCS - 1 Month | 40.35 (9.349)
  MCS - 3 Month | 48.83 (8.026)
  MCS - 6 Month | 49.99 (8.277)
  MCS - 12 Month | 50.10 (8.248)
  MCS - 18 Month | 50.48 (8.794)
  MCS - 24 Month | 48.02 (9.739)

9. Secondary Outcome: Surgical Procedure Time as Measured From Incision to Closure
Description: Surgical procedure time as measured from incision to closure (skin to skin)
Time Frame: During Procedure, up to 243 minutes
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Phasix™ ST
Number analyzed (Participants) | 120
Minutes | 85.9 (43.03)

10. Secondary Outcome: Length of Hospital Stay
Description: Number of days admitted to the hospital for index surgery
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Phasix™ ST
Number analyzed (Participants) | 120
days | 1.0 (1.35)

ADVERSE EVENTS:
Time Frame: 24 Months
Description: In this study, an Adverse Event (AE) is defined as any undesirable clinical event occurring in the abdominal space including the lower abdominal, inguinal and pubic regions (including the skin), as well as any other undesirable clinical events judged to be related to the study device or surgical procedure regardless of anatomical region. The definition of Serious AE does not deviate.
  Monitors have actively reviewed the subjects' medical records for Adverse Events during monitor visits.
Arm/Group | Phasix™ ST
All-Cause Mortality (participants affected / at risk) | 2/120
Serious Adverse Events (participants affected / at risk) | 44/120
Other Adverse Events (participants affected / at risk) | 64/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phasix™ ST (N=120)
Atrioventricular block complete (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Pseudocholinesterase deficiency (Congenital, familial and genetic disorders) | 1 (1)
Abdominal adhesions (Gastrointestinal disorders) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 1 (1)
Cyclic vomiting syndrome (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Death (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1)
Incisional Hernia (Injury, poisoning and procedural complications) | 22 (22)
Intentional Overdose (Injury, poisoning and procedural complications) | 1 (1)
Joint Injury (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 4 (4)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2)
Rib Fracture (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Ulnar neuritis (Nervous system disorders) | 1 (1)
Pelvic adhesions (Reproductive system and breast disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phasix™ ST (N=120)
Abdominal Pain (Gastrointestinal disorders) | 8 (120)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3)
Incisional hernia (Injury, poisoning and procedural complications) | 17 (17)
Procedural Pain (Injury, poisoning and procedural complications) | 17 (17)
Seroma (Injury, poisoning and procedural complications) | 9 (9)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 7 (7)
Diastasis recti abdominis (Musculoskeletal and connective tissue disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
The study was designed as a single arm observational trial without pre-defined statistical hypotheses (theories) to test; therefore, data can only be described and no treatment comparisons or conclusions can be made.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-04-16): https://cdn.clinicaltrials.gov/large-docs/98/NCT02712398/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-16): https://cdn.clinicaltrials.gov/large-docs/98/NCT02712398/SAP_001.pdf